CLINICAL TRIAL: NCT05923515
Title: A Phase I, Open, Multicenter Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of JMKX000197 Injection in the Treatment of Malignant Pleural Effusion
Brief Title: A Phase I Study of JMKX000197 Injection in the Treatment of Malignant Pleural Effusion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jemincare (Industry)
Collaborators: Zhejiang Hangyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JY-JM-0197-101
Record Dates: First submitted 2023-05-23; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- JMKX000197 Dose 1 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197
- JMKX000197 Dose 2 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197
- JMKX000197 Dose 3 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197
- JMKX000197 Dose 4 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197
- JMKX000197 Dose 5 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197
- JMKX000197 Dose 6 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197
- JMKX000197 Dose 7 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197
- JMKX000197 Dose 8 (Experimental): eight dose levels of JMKX000197 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  Interventions: Drug: JMKX000197

INTERVENTIONS:
Drug: JMKX000197 — for injection

SUMMARY:
A Phase I, Open, Multicenter Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of JMKX000197 Injection in the Treatment of Malignant Pleural Effusion

DETAILED DESCRIPTION:
Primary objectives: To evaluate the safety and tolerability of JMKX000197 injection in the treatment of patients with malignant pleural effusion, explore DLT of JMKX000197 treatment, and determine MTD and RP2D.

Secondary objectives: To evaluate the pharmacokinetic (PK)/pharmacokinetic (PD) characteristics of JMKX000197 injection in the treatment of patients with malignant pleural effusion; To evaluate preliminarily efficacy of JMKX000197 injection in patients with malignant pleural effusion; To evaluate the drug metabolic transformation of JMKX000197 injection.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined the study, signed an informed consent form, and had good compliance.
2. Age ≥ 18 years and ≤ 75 years old, regardless of gender.
3. Malignant pleural effusion confirmed by histopathology or cytopathology as moderate or above and requiring drainage (definition of moderate pleural effusion: pleural effusion ≥ 3cm in lying position by B-ultrasound, pleural effusion ≥ 4cm in sitting position by B-ultrasound, accompanied by clinical symptoms such as chest tightness, shortness of breath, and discomfort).
4. Karnofsky score ≥ 60, or physical fitness score (ECOG PS) ≤ 2.
5. Expected survival time ≥ 3 months.
6. Within 7 days before treatment, the main organ function meets the following criteria: blood routine examination criteria (without blood transfusion within 14 days): neutrophil count ≥ 1.5 × 10 ^ 9 /L, Hemoglobin ≥ 9g/dL, Platelets ≥ 100 × 10 ^ 9 /L, White blood cells ≥ 3.0 × 10 ^ 9 /L; Biochemical examination indicators should meet: total bilirubin ≤ 1.5 × ULN, ALT≤2.5 × ULT, AST≤2.5 × ULT, if accompanied by liver metastasis, ALT and AST ≤ 5 × ULN, Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate (CCr) ≥ 60ml/min; International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN.
7. No intrathoracic drug injection was performed within 1 month before signing the informed consent form, but diagnostic puncture is not excluded.
8. Women of reproductive age should agree to use contraception (such as intrauterine devices, birth control pills, or condoms) during the study period and within 6 months after the end of the study; The serum pregnancy test was negative within 7 days before enrollment and must be a non lactating patient; Men should agree to use effective contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1. Known allergies to the study drug or its excipient components.
2. The location of pleural effusion is not suitable for drainage or the patient will not benefit from intrathoracic medication (e.g., severe separation).
3. Have used interferon gene stimulating factor (STING) agonists, TNF drugs (such as Tianenfu) for thoracic injection.
4. Have participated in other clinial trials within 4 weeks before signing the informed consent form.
5. Have a history of immunodeficiency, including a positive test for human immunodeficiency virus (HIV) antibodies, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation.
6. Uncontrollable systemic infections (viruses, bacteria, fungi), including but not limited to hepatitis B surface antigen positive and hepatitis B virus DNA > 1000 IU/ml, hepatitis C virus (HCV) antibody positive or RNA positive.
7. According to the judgment of the researcher, the patient is not suitable for participating in this clinical study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | Up to approximately 7 days at each dose level
Maximum tolerated dose | Up to approximately 24 months
Recommended Phase II dose | Up to approximately 24 months

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | Up to approximately 36 days
Disease control rate, DCR | Up to approximately 36 days
Maximum observed concentration (Cmax) of JMKX000197 | Up to approximately 7 days
Time to maximum concentration (Tmax) of JMKX000197 | Up to approximately 7 days
Half-life (t1/2) of JMKX000197 | Up to approximately 7 days
Areas under the concentration-time curve from time zero extrapolated to infinity (AUC0-inf) of JMKX000197 | Up to approximately 7 days
Areas under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC0-t) of JMKX000197 | Up to approximately 7 days
Amount of Drug Excreted Via Urine and excrement During the Collection Interval 0-48 Hours Post Administration | Up to approximately 48 hours
Concentrations of IL-6 in plasma | Up to approximately 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianying Huang, Principal Investigator — Zhongnan Hospital of Wuhan University，No. 169, Donghu Road, Wuchang District, Wuhan, Hubei
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No